CLINICAL TRIAL: NCT05213559
Title: Glucose and Gastrointestinal Hormone Responses of Subjects With Overweight/Obesity After 12-week Hypocaloric Dietary Intervention Supplemented With a Cereal-based Biscuit Enriched With Plant Proteins
Brief Title: Metabolic Responses After 12-week Hypocaloric Diet Supplemented With a Cereal-based Plant Protein Biscuit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Amalia Yanni, Principal Investigator, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.14-2-2020
Record Dates: First submitted 2022-01-20; First posted 2022-01-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Appetite
Keywords: cereal-based biscuit enriched with plant proteins; appetite regulation; glycemic control; hormone responses
MeSH Terms: interventions — Plant Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wheat-based biscuit enriched with plant proteins (Experimental): Subjects follow a hypocaloric dietary intervention supplemented with certain amount of wheat-based biscuits enriched with plant proteins daily.
  Interventions: Other: wheat biscuit enriched with plant proteins
- wheat biscuit (Active Comparator): Subjects follow a hypocaloric dietary intervention supplemented with certain isocaloric amount of common wheat biscuits daily.
  Interventions: Other: common wheat biscuit

INTERVENTIONS:
Other: wheat biscuit enriched with plant proteins — Postprandial glucose and appetite-regulating hormone responses of subjects with overweight/obesity after a 12-week dietary intervention with a biscuit enriched with plant proteins
  Arms: wheat-based biscuit enriched with plant proteins
Other: common wheat biscuit — Postprandial glucose and appetite-regulating hormone responses of subjects with overweight/obesity after a 12-week dietary intervention with a common wheat biscuit
  Arms: wheat biscuit

SUMMARY:
Biscuits enjoy high popularity in the human diet and can be excellent snack alternatives and potential carriers of ingredients with appetite regulating properties. In the present study, the effects of a wheat biscuit enriched with plant proteins originated from legumes and seeds on gastrointestinal hormone responses of women with overweight/obesity after a hypocaloric dietary intervention will be examined.

DETAILED DESCRIPTION:
Women with overweight/obesity will follow a 12-week dietary intervention supplemented with a cereal-based biscuit enriched with plant proteins or a common isocaloric wheat biscuit as a daily snack.

At the beginning and at the end of the dietary intervention postprandial metabolic responses, body weight reduction and subjective appetite ratings will be examined.

ELIGIBILITY:
Inclusion Criteria:

* non-diabetic women with overweight/obesity
* constant body weight for the last three months before enrollment
* standard dietary and physical activity habits

Exclusion Criteria:

* pregnancy
* lactation
* chronic medical illness
* use of nutritional supplements
* alcohol consumption >2 drinks per day

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on gender.
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
change in postprandial glucose response | Time points: 0,30,60,91,120,180 min postprandially at week 0 and week 12.
  change in glucose iAUC and glucose concentration at certain time points at the end of the dietary intervention compared to the beginning.

SECONDARY OUTCOMES:
change in postprandial appetite regulating hormone responses | Time points: 0,30,60,91,120,180 min postprandially at week 0 and week 12.
  changes in iAUCs and concentrations at certain time points at the end of the dietary intervention compared to the beginning.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kokkinos, Professor, Study Chair — National and Kapodistrian University of Athens; Amalia Yanni, PhD, Principal Investigator — Harokopio University
Locations (1):
- Laiko General Hospital, School of Medicine, National and Kapodistrian University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No